CLINICAL TRIAL: NCT05769309
Title: Efficacy of Erector Spinae Plane Block on Postoperative Analgesia and Recovery After Off Pump Cardiac Surgery: A Randomised Trial
Brief Title: Efficacy of Erector Spinae Plane Block Analgesia After Off Pump Cardiac Surgery
Acronym: ESPB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Amal Gouda Elsayed Safan, lecturer of anaethesia, Menoufia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2/2023 ANET10-2
Record Dates: First submitted 2023-02-12; First posted 2023-03-15 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Fentanyl

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Erector spinae block group (Active Comparator): the patients will be administered bilateral Erector spinae block with 20 ml of 0.25 % bupivacaine
  Interventions: Procedure: Erector spinae block; Drug: Fentanyl
- control group (Other): no block will be done but only IV analgesia.
  Interventions: Drug: Fentanyl

INTERVENTIONS:
Procedure: Erector spinae block — After induction, the patients will be administered bilateral Erector spinae block with 20 ml of 0.25 % bupivacaine
  Arms: Erector spinae block group
Drug: Fentanyl — fentanyl boluses of 0.5-to-1 µg/kg titrated according to haemodynamic parameters.

SUMMARY:
In this study the investigators will investigate the efficacy of ESPB as a part of Enhanced recovery after surgery on postoperative analgesia and recovery criteria after off pump cardiac surgery.

DETAILED DESCRIPTION:
General anaesthesia will be induced by 0.05 mg/kg midazolam, 3 µg/kg fentanyl, 1-2mg/kg propofol, and 0.5mg/kg of Atracurium. After induction, bilateral erector spinae plane block will be performed in the block group. Intraoperative analgesia will be achieved by fentanyl boluses of 0.5-to-1 µg/kg titrated according to haemodynamic parameters. Postoperative analgesia will be managed by paracetamol 1000 mg /6hours and morphine 1-2mg boluses when pain score ≥4 1 to 2 mg to be repeated every 5 minutes if needed.

ELIGIBILITY:
Inclusion Criteria:

* age 18-70 years
* ejection fraction of > 45%
* undergoing elective off-pump cardiopulmonary bypass surgery

Exclusion Criteria:

* vertebral anomalies
* intra-aortic balloon pump in the preoperative period
* acute myocardial infarction
* local infection at the site of block
* allergy to the local anesthetic used
* morbid obesity, psychiatric disorders, neurologic deficits, alcohol and chronic opioid abuse, and patients with bleeding diathesis.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-03-22 (Actual); Primary Completion 2023-10-10 (Actual); Study Completion 2023-12-25 (Actual)

PRIMARY OUTCOMES:
Total intraoperative and postoperative opioid consumption | 48 hours
  Microgram and mg

SECONDARY OUTCOMES:
pain intensity at rest and movement | 48 hours
  numerical rating score from zero to ten ( 0=no pain, 10 =severe pain )
time to first rescue analgesia | 24hous
  minutes
Duration of mechanical ventilation | 24 hours
  hours
time to extubation | 24hours
  min
time to ambulation | 24hours
  hours
time to oral intake | 48 hours
  hours
time of chest drain removal | 5 days
  hours
time of intensive care unit stay | one week
  hours
The heart rate | 48 hours
  Beats per minutes
mean arterial blood pressure | 48 hours
  mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Islam M ElDesoky, MD, Principal Investigator — Menoufia University; AMAL G SAFAN, MD, Principal Investigator — Menoufia University; Abd-Elazeem A Elbakry, MD, Principal Investigator — Menoufia University
Locations (1):
- Menoufia university, Cairo, Shibin Elkom, Egypt

IPD SHARING:
Plan to Share IPD: No